CLINICAL TRIAL: NCT03988699
Title: Novel Tinnitus Implant System for the Treatment of Chronic Severe Tinnitus: An Early Feasibility Study
Brief Title: Novel Tinnitus Implant System for the Treatment of Chronic Severe Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew L. Carlson, M.D. (Other)
Responsible Party: Sponsor-Investigator, Matthew L. Carlson, M.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-007120
Record Dates: First submitted 2019-06-07; First posted 2019-06-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subject with severe tinnitus (Experimental): Subjects diagnosed with severe tinnitus for at least six months, and it has not responded to conventional management will have surgical implantation of the device Tinnitus Implant System.
  Interventions: Device: Tinnitus Implant System

INTERVENTIONS:
Device: Tinnitus Implant System — Device will deliver stimulation below hearing thresholds continuously or intermittently.

SUMMARY:
Researchers are gathering information on the safety and effectiveness of a novel device called the Tinnitus Implant System for the treatment of tinnitus.

DETAILED DESCRIPTION:
This study requires one year of participation with at least 21 visits to Mayo Clinic in Rochester MN for device programming and audiometric testing. The device is implanted during an outpatient surgery. Participants may keep the study device after participation is complete.

ELIGIBILITY:
Inclusion Criteria

* Age: ≥18 years of age
* Normal to moderate SNHL (≤70 dB HL; based on PTA of 0.5, 1 and 2 kHz) and WRS ≥ 75%.
* Unilateral or asymmetrical subjective tonal tinnitus
* Tinnitus present for at least 6 months, but not longer than 3 years
* Tinnitus that is disruptive

  * THI score in the severe range (≥56/100)
  * TFI score in the severe range (≥52/100)
  * Tinnitus VAS ≥50/100
* Tinnitus that is intractable, and has not been ameliorated by conventional measures such as a hearing aid or masking

Exclusion Criteria

* Age: <18 years of age
* Tinnitus present less than 6 months or longer than 3 years
* Current pregnancy
* History of brain or major ear surgery
* Prior major head trauma

  * Presence of clinically significant depressive or anxiety symptoms determined by screening using the GAD-7, PHQ-8, and SHAI

    * GAD-7 >9 (indicates clinically significant anxiety)
    * PHQ-8 >9 (indicates clinically significant depression)
    * SHAI >25 (hypochondriacal level illness anxiety)
  * Inability to assess, continue or complete trial
* Currently on antidepressants, anxiolytics or antipsychotics
* Active use of other tinnitus treatments (not including non-masking hearing aid use)
* Normal contrast-enhanced MRI of the head
* Normal temporal bone CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events | One year
  Measured by subjects meeting one or more of the following criteria: worsening bone conduction thresholds in any tested frequency (0.25, 0.5, 1, 1.5, 2, 3, or 4 kHz) from baseline by a clinically significant amount (>10 dB) or worsening in WRS from baseline by a clinically significant amount (>20%) or worsening in video head impulse test result from baseline or one or more serious AEs
Number of subjects to experience significant improvement from implantation of the device | Baseline, 3 weeks, 5 weeks, 7 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks, 13 weeks, 14 weeks, 15 weeks, 52 weeks
  Measured by subjects meeting at least two of three measurements of tinnitus severity: Tinnitus Handicap Inventory (THI) improvement by greater than 7 points using a 25-item self-assessment questionnaire with possible answers of Yes (4 points), Sometimes (2 points), and No (0 points) or Tinnitus Functional Index (TFI) improvement by greater than 13 points using a 25-item self-report questionnaire on a scale of 0 to 10 with a maximum possible score of 250 or Tinnitus visual analog scale improvement by greater than 15 points using a self-reported scale consisting of a 10 cm line with verbal descriptors (word anchors) at each end to express the extremes of the symptom; 0 mm designates no pain and 100 mm designates the greatest imaginable severity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Carlson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03988699/ICF_000.pdf